CLINICAL TRIAL: NCT00052143
Title: Prospective Huntington At Risk Observational Study (PHAROS)
Brief Title: Prospective Huntington At Risk Observational Study
Acronym: PHAROS
Status: Completed | Type: Observational
Sponsor: Huntington Study Group (Network)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01HG002449 (NIH)
Record Dates: First submitted 2003-01-23; First posted 2003-01-24 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Huntington Disease
Keywords: Huntington's disease; HD; Huntington disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to define the natural history and experiences of people who are at risk for developing Huntington's disease but who do not know their genetic status.

DETAILED DESCRIPTION:
Huntington's disease (HD) is a genetic disease characterized by changes in movement and behavior. To date, little research has been done on individuals who are at risk for developing the disease. PHAROS is an observational study designed to monitor people who are at risk for developing HD, and to survey their attitudes and beliefs about their "at-risk" status. Investigators hope this study will help answer some important questions about HD, such as: 1.) What are the earliest signs of HD and when do they start? 2.) How accurate are the measures that physicians use in detecting the onset of HD? 3.) What factors influence the age at which a person carrying the HD gene develops the illness? and 4.) In a group of people at risk for HD, how many will develop signs of the illness over a minimum three-year period of observation?

Participants in the study will be evaluated every 9 months (for 5 years) using the Unified Huntington's Disease Rating Scale (UHDRS)--a clinical tool which looks at movement, psychological and behavioral function. The participants will also be asked to complete surveys about their mood, life events, and attitudes or beliefs about being at risk for HD. A blood sample, taken at the beginning of the study, will be confidentially tested to determine if the participant has the abnormal gene for HD. Neither the participant nor any of the PHAROS physicians or coordinators will learn the results of individual gene tests.

The scientists hope that this study will provide essential information for future trials of experimental drugs for HD.

ELIGIBILITY:
Inclusion:

* Men and women between 26-55 years of age;
* Who are at risk for HD by virtue of having (or had) a parent or sibling with the illness;
* Who have never been tested for the HD gene, and who do not desire to be tested for the HD gene during the duration of the study;
* Agree to blinded (sample will be coded) genetic testing of the HD gene; and
* Who have never been diagnosed with HD.

Exclusion:

Individuals Who:

* have been diagnosed with HD;
* are taking antipsychotic medications;
* use antiemetic (anti-nausea) medications with on a regular basis (greater than 3 times per month); or
* exhibit clinical signs/symptoms of psychosis at the screening visit

Ages: 26 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: HD Community
Sampling Method: Non-Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 1999-07-09 (Actual); Primary Completion 2009-12-17 (Actual); Study Completion 2009-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Shoulson, M.D., Principal Investigator — University of Rochester
Locations (42):
- United States (37):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California at San Diego, La Jolla, California
  - UCLA School of Medicine, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - Colorado Neurological Institute, Englewood, Colorado
  - University of Connecticut, Hartford, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Hereditary Neurological Disease Center, Wichita, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Maryland at Baltimore, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - UMDNJ Huntington Disease Service Center, Stratford, New Jersey
  - Albany Medical College, Albany, New York
  - North Shore-LIJ Health System, Manhasset, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - NeuroHealth Parkinson's Disease Movement Disorders Center, Pawtucket, Rhode Island
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington and VA Puget Sound, Seattle, Washington
  - Medical College of Wisconsin-Milwaukee, Milwaukee, Wisconsin
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - The Centre for Addiction and Mental Health, Markham, Ontario
  - Hotel-Dieu Hospital-CHUM, Montreal, Quebec

REFERENCES:
- [Background] Huntington Study Group PHAROS Investigators. At risk for Huntington disease: The PHAROS (Prospective Huntington At Risk Observational Study) cohort enrolled. Arch Neurol. 2006 Jul;63(7):991-6. doi: 10.1001/archneur.63.7.991. PMID 16831969
- [Derived] Oster E, Dorsey ER, Bausch J, Shinaman A, Kayson E, Oakes D, Shoulson I, Quaid K; Huntington Study Group PHAROS Investigators. Fear of health insurance loss among individuals at risk for Huntington disease. Am J Med Genet A. 2008 Aug 15;146A(16):2070-7. doi: 10.1002/ajmg.a.32422. PMID 18627059
- See also: study website — http://www.huntington-study-group.org